CLINICAL TRIAL: NCT03239678
Title: Safe Time for Apnea After Preoxygenation With Different Oxygen Concentration During the Induction of General Anesthesia
Brief Title: Safe Time for Apnea After Preoxygenation
Acronym: STAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zijia Li, Principal Investigator, Department of anesthesiology, Sixth Affiliated Hospital, Sun Yat-sen University, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2017ZSLYEC-022
Record Dates: First submitted 2017-07-30; First posted 2017-08-04 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Anesthesia, General
Keywords: Preoxygenation; Oxygen Concentration
MeSH Terms: interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- group A (Active Comparator): 100% Oxygen
  Interventions: Drug: 100% Oxygen
- group B (Experimental): 30% Oxygen.
  Interventions: Drug: 30% Oxygen
- group C (Experimental): 21% Oxygen
  Interventions: Drug: 21% Oxygen
- group D (Experimental): 40% Oxygen
  Interventions: Drug: 40% Oxygen
- group E (Experimental): 60% Oxygen
  Interventions: Drug: 60% Oxygen
- group F (Experimental): 80% Oxygen
  Interventions: Drug: 80% Oxygen

INTERVENTIONS:
Drug: 100% Oxygen — Conventional preoxygenation with 100% oxygen
  Other Names: 100% O2
  Arms: group A
Drug: 30% Oxygen — preoxygenation with 30% oxygen
  Other Names: 30% O2
  Arms: group B
Drug: 21% Oxygen — preoxygenation with 21% oxygen
  Other Names: 21% O2
  Arms: group C
Drug: 40% Oxygen — preoxygenation with 40% oxygen
  Other Names: 40% O2
  Arms: group D
Drug: 60% Oxygen — preoxygenation with 60% oxygen
  Other Names: 60% O2
  Arms: group E
Drug: 80% Oxygen — preoxygenation with 80% oxygen
  Other Names: 80% O2
  Arms: group F

SUMMARY:
The use of 100% oxygen during the induction of general anesthesia is always preferable to have enough time to secure the airway by endotracheal intubation, because preoxygenation with a low oxygen concentration may reduce the safe time for apnea. However, using a low oxygen concentration during preoxygenation might prevent the formation of atelectasis. There is still no clear conclusion about the best oxygen concentration for preoxygenation. Our study is designed to evaluate the safety of preoxygenation with 80%, 60%, 40%, 30% and 21% oxygen by the safe time for apnea during the induction of general anesthesia.

DETAILED DESCRIPTION:
We decide to add 3 groups (80%, 60%, and 40% oxygen) in our study to fully evaluate the safety of preoxygenation with different oxygen concentration.

Zijia Li 2018.3.2

ELIGIBILITY:
Inclusion Criteria:

* Nonsmoking patients aged 18 years to 60 years
* Undergoing general anesthesia for elective surgery
* Pulse oxygen saturation ≥95% when breathing air quietly in bed
* American Society of Anesthesiologists(ASA) physical status class I-II
* Informed consent can be obtained

Exclusion Criteria:

* A suspected difficult airway
* Be allergic to midazolam, propofol , fentanyl or Cisatracurium
* Severe disease of respiratory system or cardiovascular system,or obstruction of the digestive tract
* Oxygen reserve is suspected low,or patient who does not tolerate hypoxemia well
* A history of mental disorder or patient who can not collaborate well
* Body mass index more than 30 kg/㎡

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Safe time for apnea | 10 min
  Time when peripheral oxygen saturation (SpO2) is ≥ 90% after preoxygenation.

SECONDARY OUTCOMES:
Time needed for endotracheal intubation | 1 min
  Time from when the laryngoscope blade first passes the lips to when the cuff of tracheal tube is inflated.

CONTACTS AND LOCATIONS:
Overall Officials: Sanqing Jin, MD, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University; Zijia Li, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Department of Anesthesia ,the Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lundquist H, Hedenstierna G, Strandberg A, Tokics L, Brismar B. CT-assessment of dependent lung densities in man during general anaesthesia. Acta Radiol. 1995 Nov;36(6):626-32. PMID 8519574
- [Background] Rothen HU, Sporre B, Engberg G, Wegenius G, Reber A, Hedenstierna G. Prevention of atelectasis during general anaesthesia. Lancet. 1995 Jun 3;345(8962):1387-91. doi: 10.1016/s0140-6736(95)92595-3. PMID 7760608
- [Background] Edmark L, Kostova-Aherdan K, Enlund M, Hedenstierna G. Optimal oxygen concentration during induction of general anesthesia. Anesthesiology. 2003 Jan;98(1):28-33. doi: 10.1097/00000542-200301000-00008. PMID 12502975